CLINICAL TRIAL: NCT03723980
Title: Effect of Propolis Paste as Intracanal Medicament on Post-Endodontic Pain: a Double-Blind Randomized Clinical Trial.
Brief Title: Role of Propolis Paste in Preventing Pain After Root Canal Treatment.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Juzer Shabbir Saifee (Other)
Collaborators: Dow University of Health Sciences (Other)
Responsible Party: Sponsor-Investigator, Juzer Shabbir Saifee, Principal Investigator, Dow University of Health Sciences
Organization: Dow University of Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MDSJUZER; ISRCTN66816132 (Registry Identifier: SPRINGER NATURE)
Record Dates: First submitted 2018-10-23; First posted 2018-10-30 (Actual); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-03

CONDITIONS: Pain, Postoperative
Keywords: Flare up
MeSH Terms: conditions — Pain, Postoperative | interventions — Propolis; Calcium Hydroxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group or Group I or Calcium hydroxide Group (Active Comparator)
  Interventions: Drug: Calcium Hydroxide
- Experimental Group or Group II or Propolis Group (Experimental)
  Interventions: Drug: Propolis

INTERVENTIONS:
Drug: Propolis — it is a natural product obtained from beehive. it has been evaluated for biocompatibility and toxicity; and it is found that it is extremely biocompatible material. In our study, propolis powder will be mixed with saline in a ratio of 1 : 1.5 (propolis powder(wt) / saline(vol)) to form paste; and inserted into the root canals. it will be inserted once and will remain in root canals for 4 days.
  Other Names: Bee glue
  Arms: Experimental Group or Group II or Propolis Group
Drug: Calcium Hydroxide — it is a synthetic antimicrobial intracanal medicament and gold standard to which other medicaments are being compared. approximately 150 mg of calcium hydroxide paste will be inserted in the root canal. it will be inserted only once and will remain in root canals for 4 days.
  Arms: Control Group or Group I or Calcium hydroxide Group

SUMMARY:
This study evaluates the role of propolis paste as compared to calcium hydroxide (when used as intracanal medication) in prevention and treatment of pain after root canal treatment in necrotic (infected) teeth. Half of the participants will receive calcium hydroxide, while the other half will receive propolis.

DETAILED DESCRIPTION:
Propolis is a developing herbal medicament used in various aspects on dentistry. it is extremely biocompatible; has flavanoids; which acts as anti-inflammatory and antimicrobial components.

Calcium hydroxide is a synthetic medication which is antibacterial

ELIGIBILITY:
Inclusion Criteria:

* Single rooted Necrotic teeth with symptomatic or asymptomatic periapical periodontitis having periapical widening or radiolucency without bone expansion (PAI index 2, 3 and 4).
* Teeth with favorable root morphology.
* Teeth with closed apex.

Exclusion Criteria:

* Teeth with PAI index 1 and 5.
* Patients who are on antibiotics.
* Patient with recent trauma to the jaw.
* Teeth with open apex
* Multi-rooted teeth.
* Vital teeth.
* Non-restorable teeth.
* Unfavorable root morphology (severely curved, dilacerated, severely sclerosed or obliterated).
* Teeth associated with soft tissue abscess or swelling.
* Teeth with external or internal root resorption
* Re-treatment cases.
* Periodontally compromised teeth (like mobile teeth and teeth with excessive bone loss).
* Teeth requiring endodontic surgery.
* Teeth requiring non-surgical endodontic treatment of multiple teeth in the same or opposing quadrant.
* Medically compromised patients (ASA-III and above), patients with special communication needs or who doesn't understand Urdu or English language.
* Patients allergic to bee pollen or honey products.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juzer S Saifee, Principal Investigator — Dow University of Health Sciences; Fazal R Qazi, Study Director — Dow University of Health Sciences
Locations (1):
- Dow International Dental College, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Start of recruitment : 1st october 2017 End of Recruitment: 24th april 2018
  location: Pakistan; Karachi; Dow-International dental college, Operative Dentistry; out-patient department.
Period: Overall Study
Arm/Group | Control Group or Group I or Calcium Hydroxide Group | Experimental Group or Group II or Propolis Group
Started | 40 | 40
Completed | 33 | 35
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group or Group I or Calcium Hydroxide Group | Experimental Group or Group II or Propolis Group | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (6.3) | 33.2 (6) | 33.4 (6.1)
Age, Customized [Count of Participants; unit: Participants]
  Age Range: 20 to 24 | 4 | 4 | 8
  Age Range: 25 to 29 | 7 | 4 | 11
  Age Range: 30 to 34 | 6 | 13 | 19
  Age Range: 35 to 40 | 23 | 19 | 42
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 22 | 50
  Male | 12 | 18 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 40 | 40 | 80
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Number of participants]
  Pakistan | 40 | 40 | 80
Pre-operative pain score from 0 (no pain) to 100 (worst pain) on Visual Analogue Scale [Mean (Standard Deviation); unit: units on a scale] | 13.1 (17.4) | 18.1 (12.4) | 15.6 (17.5)
Type of single-rooted teeth [Number; unit: Number of teeth]
  Maxillary Central Incisor | 4 | 2 | 6
  Maxillary Lateral Incisor | 4 | 4 | 8
  Maxillary Canine | 8 | 7 | 15
  Maxillary Second Premolar | 6 | 14 | 20
  Mandibular Lateral Incisor | 3 | 0 | 3
  Mandibular Canine | 1 | 2 | 3
  Mandibular First Premolar | 4 | 5 | 9
  Mandibular Second Premolar | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Measure: Visual Analogue Pain Scale
Description: Self recorded pain intensity by the patients at 4 hours, 12 hours, day 2, day 3 and day 4 after root canal preparation and intracanal medicament insertion (first visit). Pain intensity recorded on a Visual Analogue Scale from 0 to 100. Patients who experience no or mild pain; and do not require analgesic will record their pain intensity from 0 to 24. Patients who experience moderate pain; and require Over-the-counter analgesic will record pain intensity from 25 to 49. Patients who experience severe pain; and require use of codeine containing medicine will record their pain intensity from 50 to 74. Patients who experience extreme pain, and no medicine is able to relieve their pain will record pain intensity from 75 to 100.
  lower pain score (intensity) is a better outcome as compared to higher pain intensity (score)
Time Frame: 4 hours, 12 hours, day 2, day 3 and day 4
Population: Out of 80 patients, 12 did not return for follow-up; and no contact could be established with them. Out of these 12 patients, 7 belong to control group and 5 belong to experimental group. Hence, 33 patients in control group and 35 patients in experimental group could be analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group or Group I or Calcium Hydroxide Group | Experimental Group or Group II or Propolis Group
Number analyzed (Participants) | 33 | 35
score on a scale
  4 hours | 11.8 (18.7) | 8.8 (11.1)
  12 hours | 9.4 (16.7) | 10.3 (13.3)
  Day 2 | 3.5 (7.7) | 5.1 (9.2)
  Day 3 | 2.6 (6.4) | 3.4 (6.8)
  Day 4 | 1.9 (4.7) | 2.7 (7.3)
Statistical Analysis 1: Comparison: Control Group or Group I or Calcium Hydroxide Group vs Experimental Group or Group II or Propolis Group; Test type: Superiority; p = 0.329, ANOVA — the calculated p value is for time interval of 4 hours threshold for statistical significance= <0.05; For multiple comparisons between groups, post hoc (LSD) was applied; Mean Difference (Net) = 2.96
Statistical Analysis 2: Comparison: Control Group or Group I or Calcium Hydroxide Group vs Experimental Group or Group II or Propolis Group; Test type: Superiority; p = 0.764, ANOVA — The calculated p value is for time interval of 12 hours threshold for statistical significance= <0.05; Mean Difference (Net) = -0.92
Statistical Analysis 3: Comparison: Control Group or Group I or Calcium Hydroxide Group vs Experimental Group or Group II or Propolis Group; Test type: Superiority; p = 0.605, ANOVA — The calculated p value is for time interval of day 2 threshold for statistical significance= <0.05; Mean Difference (Net) = -1.57
Statistical Analysis 4: Comparison: Control Group or Group I or Calcium Hydroxide Group vs Experimental Group or Group II or Propolis Group; Test type: Superiority; p = 0.786, ANOVA — The calculated p value is for time interval of day 3 threshold for statistical significance= <0.05; Mean Difference (Net) = -0.82
Statistical Analysis 5: Comparison: Control Group or Group I or Calcium Hydroxide Group vs Experimental Group or Group II or Propolis Group; Test type: Superiority; p = 0.813, ANOVA — The calculated p value is for time interval of day 4 threshold for statistical significance= <0.05; Mean Difference (Net) = -0.72

2. Secondary Outcome: Acute Increase in Pain Score (Acute Exacerbation of Pain)
Description: An increase of 20 or more points on Visual Analogue Pain Scale from pain score of previous time interval
  Information about the Visual Analogue Scale:
  * it consists of pain score from 0 to 100.
  * The higher the pain score; the worse the pain
  * An increase of a total of at least 20 pain score points from previous pain score reading indicate that pain has increased significantly and will be reported as "flare-up"
Time Frame: 4 hours, 12 hours, day 2, day 3, and day 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group or Group I or Calcium Hydroxide Group | Experimental Group or Group II or Propolis Group
Number analyzed (Participants) | 33 | 35
Participants
  4 hours: Flare up | 4 | 1
  4 hours: No flare up | 29 | 34
  12 hours: Flare up | 0 | 4
  12 hours: No flare up | 33 | 31
  Day 2: Flare up | 0 | 1
  Day 2: No flare up | 33 | 34
  Day 3: Flare up | 0 | 0
  Day 3: No flare up | 33 | 35
  Day 4: Flare up | 0 | 0
  Day 4: No flare up | 33 | 35
  Total: Flare up | 4 | 6
  Total: No flare up | 29 | 29

3. Secondary Outcome: Difference of Pain Score Between Different Time Intervals
Description: Visual Analogue Pain Score information:
  * pain intensity is measured with this scale
  * minimum pain score reading on Visual Analogue Scale is 0 and Maximum is 100
  * higher values represent worse pain and lower values represent lesser pain
  this pain score is recorded pre-operatively, then at time intervals of 4 hours, 12 hours, day 2, day 3 and day 4.
  the comparison of mean pain scores of different time intervals will be made.
Time Frame: 4 hours, 12 hours, day 2, day 3, and day 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control Group or Group I or Calcium Hydroxide Group | Experimental Group or Group II or Propolis Group
Number analyzed (Participants) | 33 | 35
score on a scale
  Pain score difference; pre-operative - 4 hours | 2.97 (3) | 11.80 (2.9)
  Pain score difference; 4 hours - 12 hours | 2.33 (3) | -1.54 (2.9)
  Pain score difference; 12 hours - day 2 | 5.88 (3) | 5.23 (2.9)
  Pain score difference; day 2 - day 3 | 0.94 (3) | 1.69 (2.9)
  Pain score difference; day 3 - day 4 | 0.67 (3) | 0.77 (2.9)
Statistical Analysis 1: Comparison: Control Group or Group I or Calcium Hydroxide Group; Test type: Other; p = 0.334, ANOVA — The calculated p value is for the difference between pre-operative time interval and 4 hours time interval. Threshold for statistical significance= <0.05; Mean Difference (Net) = 2.97, Standard Error of Mean 3
Statistical Analysis 2: Comparison: Control Group or Group I or Calcium Hydroxide Group; Test type: Other; p = 0.448, ANOVA — The calculated p value is for the difference between time interval of 4 hours and time interval of 12 hours. Threshold for statistical significance= <0.05; Mean Difference (Net) = 2.33, Standard Error of Mean 3
Statistical Analysis 3: Comparison: Control Group or Group I or Calcium Hydroxide Group; Test type: Other; p = 0.056, ANOVA — The calculated p value is for the difference between time intervals of 12 hours and day 2 Threshold for statistical significance= <0.05; Mean Difference (Net) = 5.88, Standard Error of Mean 3
Statistical Analysis 4: Comparison: Control Group or Group I or Calcium Hydroxide Group; Test type: Other; p = 0.760, ANOVA — The calculated p value is for the difference between time intervals of day 2 and day 3 Threshold for statistical significance= <0.05; Mean Difference (Net) = 0.94, Standard Error of Mean 3
Statistical Analysis 5: Comparison: Control Group or Group I or Calcium Hydroxide Group; Test type: Other; p = 0.828, ANOVA — The calculated p value is for the difference between time intervals of day 3 and day 4 Threshold for statistical significance= <0.05; Mean Difference (Net) = 0.67, Standard Error of Mean 3
Statistical Analysis 6: Comparison: Experimental Group or Group II or Propolis Group; Test type: Other; p = 0.000, ANOVA — The calculated p value is for the difference between pre-operative time interval and 4 hours time interval Threshold for statistical significance= <0.05; Mean Difference (Net) = 11.80, Standard Error of Mean 2.9
Statistical Analysis 7: Comparison: Experimental Group or Group II or Propolis Group; Test type: Other; p = 0.605, ANOVA — The calculated p value is for the difference between time interval of 4 hours and time interval of 12 hours Threshold for statistical significance= <0.05; Mean Difference (Net) = -1.54, Standard Error of Mean 2.9
Statistical Analysis 8: Comparison: Experimental Group or Group II or Propolis Group; Test type: Other; p = 0.80, ANOVA — [p-value comment as in outcome 3, analysis 3]; Mean Difference (Net) = 5.23, Standard Error of Mean 2.9
Statistical Analysis 9: Comparison: Experimental Group or Group II or Propolis Group; Test type: Other; p = 0.574, ANOVA — [p-value comment as in outcome 3, analysis 4]; Mean Difference (Net) = 1.69, Standard Error of Mean 2.9
Statistical Analysis 10: Comparison: Experimental Group or Group II or Propolis Group; Test type: Other; p = 0.796, ANOVA — [p-value comment as in outcome 3, analysis 5]; Mean Difference (Net) = 0.77, Standard Error of Mean 2.9

4. Other Pre Specified Outcome: Difference of Pain Scores Between Males and Females
Description: Information about Visual Analogue Scale for rating pain scores:
  * minimum pain score on this scale is 0 and maximum is 100
  * more the pain score; worse the pain
  * mean pain score difference between males and females at different time intervals was assessed
  * scale is divided into 4 segments: 0 to 24 (no or mild pain), 25 to 49 (moderate pain), 50 to 74 (severe pain); 75 to 100 (extreme pain).
Time Frame: 4 hours, 12 hours, day 2, day 3, and day 4
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pain Experienced by Males: Irrespective of the medicament inserted; Pain severity based of Visual analogue scale is analyzed both quantitatively and qualitatively in males.
- Pain Experienced by Females: Irrespective of the medicament inserted; Pain severity based of Visual analogue scale is analyzed both quantitatively and qualitatively in females.
Arm/Group | Pain Experienced by Males | Pain Experienced by Females
Number analyzed (Participants) | 25 | 43
score on a scale
  4 hours | 9.8 (11.9) | 10.4 (16.9)
  12 hours | 11.6 (14.5) | 8.8 (15.2)
  Day 2 | 7.8 (11) | 2.3 (5.8)
  Day 3 | 5.8 (8.9) | 1.40 (4)
  Day 4 | 5 (9.2) | 0.70 (2.1)
Statistical Analysis 1: Comparison: Pain Experienced by Males vs Pain Experienced by Females; Test type: Other; p = 0.412, Wilcoxon (Mann-Whitney) — The p-value calculated is for pain score difference at 4 hours Threshold for statistical significance= <0.05; Mean Difference (Net) = -0.6
Statistical Analysis 2: Comparison: Pain Experienced by Males vs Pain Experienced by Females; Test type: Other; p = 0.94, Wilcoxon (Mann-Whitney) — The p-value calculated is for pain score difference at 12 hours Threshold for statistical significance= <0.05; Mean Difference (Net) = 2.8
Statistical Analysis 3: Comparison: Pain Experienced by Males vs Pain Experienced by Females; Test type: Other; p = 0.035, Wilcoxon (Mann-Whitney) — The p-value calculated is for pain score difference at Day 2 Threshold for statistical significance= <0.05; Mean Difference (Net) = 5.5
Statistical Analysis 4: Comparison: Pain Experienced by Males vs Pain Experienced by Females; Test type: Other; p = 0.023, Wilcoxon (Mann-Whitney) — The p-value calculated is for pain score difference at Day 3 Threshold for statistical significance= <0.05; Mean Difference (Net) = 4.4
Statistical Analysis 5: Comparison: Pain Experienced by Males vs Pain Experienced by Females; Test type: Other; p = 0.020, Wilcoxon (Mann-Whitney) — The p-value calculated is for pain score difference at Day 4. Threshold for statistical significance= <0.05; Median Difference (Net) = 4.3

5. Other Pre Specified Outcome: Difference of Pain Scores Between Different Age Groups
Description: Information about Visual Analogue Scale for rating pain scores:
  * minimum pain score on this scale is 0 and maximum is 100
  * more the pain score; worse the pain
  * mean pain score difference between different age groups: 20 to 24; 25 to 29; 30 to 34; and 35 to 40 at different time intervals was assessed
  * scale is divided into 4 segments: 0 to 24 (no or mild pain), 25 to 49 (moderate pain), 50 to 74 (severe pain); 75 to 100 (extreme pain).
Time Frame: 4 hours, 12 hours, day 2, day 3, and day 4
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Age Group; 20 to 24: For ease of tabulating results; patients were distributed in 4 groups according to their age: 20 to 24; 25 to 29; 30 to 34; 35 to 40
  This age group consisted of total number of 6 patients. 3 belonged to control group and 3 belonged to experimental group
- Age Group; 25 to 29: For ease of tabulating results; patients were distributed in 4 groups according to their age: 20 to 24; 25 to 29; 30 to 34; 35 to 40
  This age group consisted of total number of 10 patients. 6 belonged to control group and 4 belonged to experimental group
- Age Group; 30 to 34: For ease of tabulating results; patients were distributed in 4 groups according to their age: 20 to 24; 25 to 29; 30 to 34; 35 to 40
  This age group consisted of total number of 17 patients. 6 belonged to control group and 11 belonged to experimental group
- Age Group; 35 to 40: For ease of tabulating results; patients were distributed in 4 groups according to their age: 20 to 24; 25 to 29; 30 to 34; 35 to 40
  This age group consisted of total number of 35 patients. 18 belonged to control group and 17 belonged to experimental group
Arm/Group | Age Group; 20 to 24 | Age Group; 25 to 29 | Age Group; 30 to 34 | Age Group; 35 to 40
Number analyzed (Participants) | 6 | 10 | 17 | 35
score on a scale
  Mean pain score; 4 hours | 7.1 (9.1) | 14.5 (15.1) | 14.6 (21.2) | 7.4 (12.1)
  Mean pain score; 12 hours | 8.3 (14.3) | 12.9 (17.9) | 13.6 (16.3) | 7.4 (13.5)
  Mean pain score; day 2 | 0 (0) | 10.6 (13.1) | 3.7 (6.9) | 3.6 (7.7)
  Mean pain score; day 3 | 1.5 (3.6) | 4 (9.6) | 1.5 (4.2) | 3.7 (6.9)
  Mean pain score; day 4 | 0 (0) | 2.1 (6.2) | 0.3 (1.2) | 3.7 (7.6)
Statistical Analysis 1: Comparison: Age Group; 20 to 24 vs Age Group; 25 to 29 vs Age Group; 30 to 34 vs Age Group; 35 to 40; Test type: Other; p = 0.15, Kruskal-Wallis — The p-value calculated is for pain score difference at 4 hours Threshold for statistical significance= <0.05
Statistical Analysis 2: Comparison: Age Group; 20 to 24 vs Age Group; 25 to 29 vs Age Group; 30 to 34 vs Age Group; 35 to 40; Test type: Other; p = 0.36, Kruskal-Wallis — The p-value calculated is for pain score difference at 12 hours Threshold for statistical significance= <0.05
Statistical Analysis 3: Comparison: Age Group; 20 to 24 vs Age Group; 25 to 29 vs Age Group; 30 to 34 vs Age Group; 35 to 40; Test type: Other; p = 0.13, Kruskal-Wallis — The p-value calculated is for pain score difference at day 2 Threshold for statistical significance= <0.05
Statistical Analysis 4: Comparison: Age Group; 20 to 24 vs Age Group; 25 to 29 vs Age Group; 30 to 34 vs Age Group; 35 to 40; Test type: Other; p = 0.55, Kruskal-Wallis — The p-value calculated is for pain score difference at day 3 Threshold for statistical significance= <0.05
Statistical Analysis 5: Comparison: Age Group; 20 to 24 vs Age Group; 25 to 29 vs Age Group; 30 to 34 vs Age Group; 35 to 40; Test type: Other; p = 0.17, Kruskal-Wallis — The p-value calculated is for pain score difference at day 4 Threshold for statistical significance= <0.05

ADVERSE EVENTS:
Time Frame: 4 hours, 12 hours, day 2, day 3, and day 4
Arm/Group | Control Group or Group I or Calcium Hydroxide Group | Experimental Group or Group II or Propolis Group
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 4/40 | 6/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group or Group I or Calcium Hydroxide Group (N=40) | Experimental Group or Group II or Propolis Group (N=40)
Flare-up (General disorders) | 4 | 6 — Increase of 20 or more pain score points from pain score of previous time interval on Visual Analogue Scale

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/80/NCT03723980/Prot_SAP_ICF_000.pdf